CLINICAL TRIAL: NCT03246581
Title: Protocol With Amendments 1 and 2: Phase I Randomised, Two-period 21 Day Crossover Study in Healthy Male and Female Volunteers to Compare the Steadystate Pharmacokinetics of Tiotropium Delivered From a Test pMDI Product With Spiriva Respimat
Brief Title: Two-period 21 Day Cross-over Study to Compare the Pharmacokinetics of Tiotropium From Two Inhalers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kindeva Drug Delivery (Industry)
Collaborators: Simbec Research (Industry); 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CSP-07-000040
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: inhalation; anticholinergic
MeSH Terms: conditions — Respiratory Aspiration | interventions — Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): tiotropium pMDI 2 inhalations
  Interventions: Drug: Tiotropium
- Commercial Product (Active Comparator): tiotropium pMDI 2 inhalations
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium — inhalation
  Other Names: Spiriva Respimat

SUMMARY:
The purpose of this study is to compare the absorption of a test inhalation product with the reference product in healthy volunteers.

DETAILED DESCRIPTION:
Healthy subjects will be enrolled and will receive doses of a test inhalation product and a reference inhalation product for 28 days according to a crossover design. Plasma tiotropium levels will be measured predose and over 24 hours postdose on days 1 and 28.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer
* Willing and able to give informed consent
* Willing to withhold all alcoholic beverages for 48 hours and all xanthine- containing foods and beverages for 24 hours prior to reporting to clinic
* Subjects must agree to use an adequate method of contraception from admission through 12 weeks after last administration

Exclusion Criteria:

* Evidence or history of clinically significant abnormalities or disease or chronic respiratory disorders
* Any presence or history of a clinically significant allergy including any adverse reaction to study drug
* History of drug or alcohol abuse within the past 2 years
* Smoked tobacco within the past 6 months or have a history of more than 10- pack years (number of packs smoked per day x number of years smoked)
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Have received any prescription medication within 4 weeks or investigational medication within 12 weeks of study (exception: contraceptives are permitted)
* Have received any non-prescription medication within 14 days prior to dosing (exception: paracetamol use within 2 days)
* Upper respiratory tract infection (excluding otitis media) within 14 days of the first study day, or lower respiratory tract infection within the last 3 months
* If female, nursing, lactating or pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-01-21 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 24 hours
  noncompartmental analysis

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Sessions, PhD, Study Chair — 3M
Locations (1):
- 3M Health Care, Loughborough, United Kingdom